CLINICAL TRIAL: NCT05798338
Title: Characterization of Extracellular Vesicles in Breast Cancer Patients' Plasma by Single Molecule Detection Array (SiMoA) Digital ELISA
Brief Title: Characterization of Extracellular Vesicles in Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Fabio Corsi, Prof, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2490
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early Breast Cancer patients: * Diagnosis of early breast cancer;
  * Indication for surgery after multidisciplinary discussion.
  Interventions: Diagnostic Test: Blood sample
- Metastatic Breast Cancer patients: * First diagnosis of metastatic breast cancer confirmed by cytological/histological examination or by imaging;
  * Indication to chemotherapy.
  Interventions: Diagnostic Test: Blood sample
- Healthy patients: - Patients having a negative mammography or breast ultrasound within 12 months from the study enrollment.
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Analysis of plasma in order to quantify and characterize EVs

SUMMARY:
Extracellular vesicles (EVs) are lipid bilayer-delimited particles, naturally released from cells and mediators of intercellular cross-talk. In breast cancer (BC), EVs seem to be involved in the tumor microenvironment's shaping, in cancer cells invasion and in the set-up of metastasis.

Clinical studies have provided initial evidence that these vesicles may have a prognostic and predictive value in breast cancer. Considering their ubiquitous presence in body fluids and their minimally invasive assessment through blood sampling, EVs could have a potential as liquid biopsy-derived biomarkers. Their quantification though is a complex task requiring complicated and time-consuming pre-analytical procedures of EVs isolation.

This protocol want to develop a new method for the detection of tumor-derived-EVs associated proteins, based on the use of Single Molecule Array (SiMoA), a digital ELISA technology able to detect and quantify extremely low concentrations of target proteins or particles.

The aim of this study is to evaluate how this new technology can allow the quantification of EVs plasma levels in patients affected by BC, providing useful diagnostic and prognostic information.

DETAILED DESCRIPTION:
This is a prospective, observational, monocentric and no profit study. The study involves the analysis of plasma from patients with breast cancer in order to quantify and characterize tumor-derived EVs at specific disease stages.

The enrollment of consecutive patients affected by BC referring to an EUSOMA-accredited Breast Unit is planned.

The patients will be divided into three pre-planned groups, as follows:

Population 1: patients diagnosed with early breast cancer patients (stage I-III) with indication to curative surgery.

Population 2: a control group made of sex- and age-matched healthy volunteers, not affected by cancer or chronic diseases.

Population 3: patients with metastatic breast cancer diagnosis. For each patient a blood sample will be collected and plasma will be isolated. A new SiMoA assay based on the use of anti-CD63 and anti-CD9 antibodies, two well known protein markers of EVs, will be used to capture and quantify EVs directly from plasma without requiring any prior sample processing.

The study will be conducted following the International Conference on Harmonization [ICH] Good Clinical Practice [GCP] guidelines. The Ethical Committee of ICS Maugeri authorized the study as protocol 2490/2020.

ELIGIBILITY:
Inclusion Criteria:

* Signing of a specific informed consent for participation to the study
* Female sex

Population 1:

* Diagnosis of early breast cancer;
* Indication for surgery after multidisciplinary discussion.

Population 2:

- Patients having a negative mammography or breast ultrasound within 12 months from the study enrollment.

Population 3:

* Diagnosis of metastatic breast cancer confirmed by cytological/histological examination or by imaging;
* Indication to chemotherapy.

Exclusion Criteria:

Population 1:

* Presence of distant metastases
* Synchronous presence of a different tumor
* Indication to neoadjuvant chemotherapy

Population 2:

* Diagnosis of breast cancer
* Synchronous presence of a different tumor or chronic disease

Population 3:

- Patients who are unfit for systemic chemotherapy treatment

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is gender specific
Study Population: Breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
EVs levels in early BC | 36 months
  Determination of plasma EVs levels in patients with EBC by SIMOA digital ELISA and evaluation of the difference of their concentration compared to healthy controls
EVs levels in metastatic BC | 36 months
  Determination of plasma EVs levels in patients with first diagnosis of metastatic BC by SIMOA digital ELISA and evaluation of the difference of their concentration compared to healthy controls

SECONDARY OUTCOMES:
EVs levels after surgery | 36 months
  Determination of plasma EVs levels in patients with early BC one month after surgery and comparison with pre-surgery EVs levels in order to evaluate any qualitative of quantitative modifications in circulating EVs
EVs levels after chemotherapy treatment | 36 months
  Determination of plasma EVs levels in patients with first diagnosis of metastatic BC after 4 months of systemic therapy and comparison with pre-therapy EV's plasma levels

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No